CLINICAL TRIAL: NCT04681651
Title: A Randomized Controlled Trial Assessing the Efficacy and Safety of Normobaric Hyperoxia for Acute Ischemic Stroke Patients Undergoing Endovascular Treatment
Brief Title: Normobaric Hyperoxia Combined With Endovascular Treatment in Acute Ischemic Stroke (OPENS-2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: Tianjin Huanhu Hospital (Other); Shengli Oilfield Hospital (Other); Beijing Fengtai You'anmen Hospital (Unknown); Jiujiang University Affiliated Hospital (Other Government); Zhangzhou Municipal Hospital of Fujian Province (Other); Baotou Central Hospital (Other); Luoyang Central Hospital (Other); Nanyang Central Hospital (Other); Qingdao Central Hospital (Other); The Third People's Hospital of Jinan (Unknown); Rizhao People's Hospital (Other); Anyang People's Hospital (Unknown); Shanghai 10th People's Hospital (Other); Dalian Municipal Central Hospital (Other); Zhoukou Central Hospital (Other); Nanshi Hospital of Nanyang (Unknown); The second Nanning People's Hospital (Unknown); Zhumadian Central Hospital (Other); Taizhou Hospital (Other); Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OPENS-2
Record Dates: First submitted 2020-12-06; First posted 2020-12-23 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-03

CONDITIONS: Stroke, Acute; Neuroprotection
Keywords: Normobaric hyperoxia; Endovascular treatment; Acute ischemic stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBO group (Experimental): Normobaric Hyperoxia combined with endovascular mechanical thrombectomy
  Interventions: Drug: Normobaric Hyperoxia; Procedure: Endovascular Thrombectomy
- Control group (Placebo Comparator): Inhale air placebo plus endovascular mechanical thrombectomy
  Interventions: Drug: Sham Normobaric Hyperoxia; Procedure: Endovascular Thrombectomy

INTERVENTIONS:
Drug: Normobaric Hyperoxia — Within 6 hours after stroke onset, patients were randomized into the NBO group and immediately given 100% oxygen inhalation (no more than 30 minutes after randomization) at a ventilation rate of 10L/ min using a sealed non-ventilating oxygen storage mask and keep giving oxygen for 4 hours. If the patient needs to be intubated with a ventilator to maintain ventilation, the FiO2 should be set to 1.0.
  Other Names: NBO
  Arms: NBO group
Drug: Sham Normobaric Hyperoxia — For Sham NBO group, Patients were immediately given oxygen inhalation (no more than 30 minutes after randomization) at a ventilation rate of 1l/min using the same mask and keep giving oxygen for 4 hours. If the patient needs to be intubated with a ventilator to maintain, the FiO2 should be set to 0.3 and gradualy incerased if spO2≤94%；
  Other Names: Sham NBO
  Arms: Control group
Procedure: Endovascular Thrombectomy — EVT is the international guidelines for the treatment of acute ischemic stroke with lage vessel occlusion.
  Other Names: EVT

SUMMARY:
The current endovascular treatment has increased the recanalization rate to more than 90%. Even so, the prognosis rate of stroke is still less than 50%. Our previous research confirmed that the neuroprotective effect of Normobaric Hyperoxia (NBO) from multiple perspectives. However, the clinical study on NBO was not satisfactory, which might be due to the absence of vascular recanalization therapy. Therefore, The investigators conducted this RCT study to further explore the Efficacy and safety of NBO combined with endovascular treatment in patients with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria

1. It conforms to the indications for endovascular thrombectomy
2. 18 ≦ Age ≦ 80 years old.
3. The clinical symptoms and signs are consistent with acute anterior circulation large vessel occlusion; 10≤NIHSS≤20；
4. (Level of consciousness) NIHSS score 0 or 1;
5. The time from onset to randomization is within 6 hours of onset;
6. The mRS score before stroke is 0-1;
7. Patient and family members sign informed consent. Image inclusion criteria

1. Preoperative CT or MR or DSA angiography found large vessel occlusion (internal carotid artery or middle cerebral artery M1 segment) that were consistent with symptoms and signs; 2. ASPECT score ≥ 6 points 3. <1/3 MCA area involvement (confirmed by CT or MRI)

Exclusion Criteria:

* General exclusion criteria

  1. Rapid neurological function improvement, NIHSS score less than 10 points, or evidence of vessel recanalization prior to randomization;
  2. Seizures at stroke onset;
  3. Intracranial hemorrhage;
  4. Symptoms suggestive of subarachnoid hemorrhage, even if CT scan was normal;
  5. Known hemorrhagic diathesis, coagulation factor deficiency, or on anticoagulant therapy with INR > 3.0 or PTT > 3 times normal;
  6. Platelet count of less than 100,000 per cubic millimeter;
  7. Severe hepatic or renal dysfunction;
  8. Severe, sustained hypertension (Systolic Blood Pressure >185 mmHg or Diastolic Blood Pressure >110 mmHg)
  9. Baseline blood glucose of <50mg/dL (2.78 mmol) or >400mg/dL (22.20 mmol)
  10. Active and chronic obstructive pulmonary disease or acute respiratory distress syndrome;
  11. >3 L/min oxygen required to maintain peripheral arterial oxygen saturation (SaO2) 95% as per current stroke management guidelines;
  12. Medically unstable;
  13. Life expectancy<90 days;
  14. Patients who could not complete the 90-day follow-up;
  15. Evidence of intracranial tumor;
  16. Patients with anemia or polycythemia vera or other situations that require urgent oxygen inhalation;
  17. Patients with upper gastrointestinal bleeding or nausea or vomiting so that they cannot cooperate with the mask to inhale oxygen.
  18. A history of severe allergies to contrast agents;
  19. There are any other conditions that are not suitable for endovascular treatment.

Image exclusion criteria

1. CTA/MRAshows excessive bending of blood vessels, which may hinder the delivery of the device;
2. Suspected cerebrovascular inflammation based on medical history and CTA/MRA;
3. Suspected aortic dissection based on medical history and CTA/MRA
4. CTA/MRA confirmed multi-vascular area occlusion (such as bilateral anterior circulation or anterior/posterior circulation), or bilateral infarction or multi- regional infarction;
5. CTA/MRAconfirmed moyamoya disease or moyamoya syndrome;
6. CT/MRI confirmed the obvious effect of midline shift
7. CT/MRI confirmed the presence of intracranial tumors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) score | 90 ± 14 days after randomization
  the mRs is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability, and 6=death)

SECONDARY OUTCOMES:
Cerebral infarct volume | 24-48h after randomization
  The infarct volume of cerebral infarct is evaluated by MRI or CT
The proportion of good prognosis | 90 ± 14 days after randomization
  defined by mRS 0-2
The proportion of functional independence | 90 ± 14 days after randomization
  defined by mRS 0-1
The proportion of severe disability | 90 ± 14 days after randomization
  defined by mRS 4-6
Scores assessed by National Institutes of Health Stroke Scale(NIHSS) | 24 ± 6 hours, 72 ± 24 hours, 7 ± 2 days after randomization
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits
The proportion of neurological function improvement | 24 ± 6 hours after randomization
  ≥ 4 point reduction in NIHSS score from baseline
Successful vessel recanalization | Immediately after procedure
  Successful vessel recanalization is defined by eTICI 2b/2c/3 on final angiogram. Extended treatment in cerebral ischaemia (eTICI) score range from 0 to 3, with higher scores indicating better reperfusion
Vessel recanalization | 24 ± 6 hours after randomization
  Vessel recanalization is evaluated by CTA or MRA and assessed by AOL grades. Arterial Occlusive Lesion (AOL) range from 0 to 3, with higher scores indicating better recanalization
Arterial oxygen partial pressure | after 4 hours of oxygen therapy
  Laboratory indicators, obtained by arterial blood gas analysis
Barthel Index (BI) | 90 ± 14 days after randomization
  the BI is an ordinal disability score of 10 categories (range from 0 to 100, higher values indicate better prognosis)
EuroQol five dimensions questionnaire（EQ-5D） | 90 ± 14 days after randomization
  The score ranges from 0 to 100, with higher scores indicating optimal health
Days of hospitalization | 90 ± 14 days after randomization
  Length of stay in hospital
All-cause mortality | 90 ± 14 days after randomization
  Safety endpoint; the proportion of all patients who died in each group
Serious adverse events | 90 ± 14 days after randomization
  Safety endpoint; the proportion of serious adverse events in each group
Stroke-related mortality | 90 ± 14 days after randomization
  Safety endpoint; the proportion of stroke related deaths in each group
Oxygen-related adverse events | 90 ± 14 days after randomization
  Safety endpoint; the proportion of oxygen-related adverse events in each group, including severe lung infection, pneumothorax, atelectasis, respiratory failure, acute respiratory distress syndrome, and cardiopulmonary arrest
Adverse events of special interest | 90 ± 14 days after randomization
  Safety endpoint; the proportion of adverse events of special interest in each group, including malignant brain edema, perioperative myocardial infarction, and acute heart failure
Symptomatic intracranial hemorrhage | 24 ± 6 hours after randomization
  Safety endpoint; according to ECASS II definition
Any intracranial hemorrhage | 24 ± 6 hours after randomization
  Safety endpoint; the proportion of any intracranial hemorrhage in each group
Early neurological deterioration (END) | 24 ± 6 hours after randomization
  Safety endpoint; defined as ≥4 point increase in NIHSS score from baseline
Systolic and diastolic blood pressure | 24 ± 6 hours after randomization
  Safety endpoint; vital signs
Heart rate | 24 ± 6 hours after randomization
  Safety endpoint; vital signs
Respiratory rate | 24 ± 6 hours after randomization
  Safety endpoint; vital signs
Oxygen saturation | 24 ± 6 hours after randomization
  Safety endpoint; vital signs
PH of arterial blood gas analysis | after 4 hours of oxygen therapy
  Safety endpoint
PaCO2 of arterial blood gas analysis | after 4 hours of oxygen therapy
  Safety endpoint
Lactic acid of arterial blood gas analysis | after 4 hours of oxygen therapy
  Safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD,PhD, Principal Investigator — Capital Medical University
Locations (1):
- Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Li W, Lan J, Wei M, Liu L, Hou C, Qi Z, Li C, Jiao L, Yang Q, Chen W, Liu S, Yue X, Dong Q, Yuan H, Gao Z, Wu X, Wen C, Li T, Jiang C, Li D, Chen Z, Shi J, Shi W, Yuan J, Qin Y, Li B, Fisher M, Feng W, Liu KJ, Ji X; OPENS-2 Investigators. Normobaric hyperoxia combined with endovascular treatment for acute ischaemic stroke in China (OPENS-2 trial): a multicentre, randomised, single-blind, sham-controlled trial. Lancet. 2025 Feb 8;405(10477):486-497. doi: 10.1016/S0140-6736(24)02809-5. PMID 39922675